CLINICAL TRIAL: NCT06287177
Title: Multicenter Study on the Evaluation of Adherence, Persistence and Efficacy of Treatment With Inclisiran in Italy - CHOLINET (CHOLesterol Italian Inclisiran NETwork)
Brief Title: Multicenter Study on the Evaluation of Adherence, Persistence and Efficacy of Treatment With Inclisiran in Italy
Acronym: CHOLINET
Status: Recruiting | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Pasquale Perrone Filardi, Professor, Federico II University
Other Study IDs: Protocol 28/2023
Record Dates: First submitted 2024-02-20; First posted 2024-02-29 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — ALN-PCS

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Subjects with hyperlipidaemia under Inclisiran treatment
  Interventions: Drug: Inclisiran

INTERVENTIONS:
Drug: Inclisiran — Injection

SUMMARY:
Evaluation of adherence, persistence and efficacy of treatment with Inclisiran in a real-life Italian population

ELIGIBILITY:
Inclusion Criteria:

* Patients under Inclisiran treatment

Exclusion Criteria:

* Age < 18 years o > 80 years
* Patients who refuse to participate and to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes patients from Italy, who have received Inclisiran as part of routine clinical management of their hyperlipidaemia, based on national reimbursement criteria, at time of enrollment
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2030-11-01 (Estimated)

PRIMARY OUTCOMES:
Description of adherence to treatment with Inclisiran in a real-life Italian population | at 3 months and every 6 months thereafter
  Adherence will be assessed in terms of Medical Possession Ratio (MPR) which is defined as the ratio between the treatment units dispensed during the treatment period and the duration of the treatment period itself.
Description of persistence to treatment with Inclisiran in a real-life Italian population | at 3 months and every 6 months thereafter
  Persistence will be assessed in terms of therapeutic continuity from the start of treatment to enrollment.
Description of efficacy of treatment with Inclisiran in a real-life Italian population | at 3 months and every 6 months thereafter
  Efficacy of treatment will be evaluated as a change in the LDL (deltaLDL) value from the start of treatment (percentage and absolute value). The deltaLDL will be calculated as an overall (mean and median value), by type of prevention (primary and secondary), by type of basic therapy, by demographic variables (age, sex, geographic origin, basal LDL levels) and by type of prescriber (hospital or territorial).

CONTACTS AND LOCATIONS:
Locations (1):
- Federico II University of Naples, Department of Advanced Biomedical Sciences, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No